CLINICAL TRIAL: NCT03697655
Title: Pre-emptive Daratumumab Therapy of Minimal Residual Disease Reappearance or Biochemical Relapse in Multiple Myeloma (PREDATOR)
Brief Title: Pre-emptive Daratumumab Therapy of Minimal Residual Disease Reappearance or Biochemical Relapse in Multiple Myeloma
Acronym: PREDATOR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Polish Myeloma Consortium (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Bioscience, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PMC008
Record Dates: First submitted 2018-09-20; First posted 2018-10-05 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: treatment arm and control (observation) arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PREDATOR-BR Cohort A (Experimental): n=46, Daratumumab 20 MG/ML [Darzalex], 16 mg/kg body weight administered as an intravenous infusion
  Interventions: Drug: Daratumumab 20 MG/ML [Darzalex]
- PREDATOR-BR Cohort B (No Intervention): n=46, Control Group, Observation (no treatment)
- PREDATOR-MRD Cohort A (Experimental): n=59, Daratumumab 20 MG/ML [Darzalex], 16 mg/kg body weight administered as an intravenous infusion
  Interventions: Drug: Daratumumab 20 MG/ML [Darzalex]
- PREDATOR-MRD Cohort B (No Intervention): n=59, Control Group, Observation (no treatment)

INTERVENTIONS:
Drug: Daratumumab 20 MG/ML [Darzalex] — Daratumumab dose 16 mg/kg body weight to be administered as an IV infusion. treatment given until clinical progression or SPR but no longer than 73 weeks
  Other Names: Darzalex
  Arms: PREDATOR-BR Cohort A; PREDATOR-MRD Cohort A

SUMMARY:
PREDATOR is a study investigating a role of preemptive daratumumab therapy for preclinical relapse or progression of multiple myeloma (MM).

DETAILED DESCRIPTION:
The study is composed of two phase 2 randomized multi-center substudies:

* PREDATOR-BR: to investigate the role of daratumumab in the setting of biochemical relapse
* PREDATOR-MRD: to investigate the role of daratumumab in minimal residual disease (MRD) reappearance

ELIGIBILITY:
PREDATOR-BR:

Inclusion Criteria:

1. Patients with diagnosed symptomatic MM who have completed one or two prior lines of therapy; single or tandem autologous stem cell transplant is not considered a separate line of therapy and is not mandatory; and have achieved at least PR to last line of therapy, and who experience asymptomatic biochemical progression not meeting criteria for SPR.
2. Males and females ≥18 years of age.
3. Life expectancy of more than 3 months.
4. ECOG performance status of 0-2.
5. Adequate hepatic function, with bilirubin ≤1.5 x ULN and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN.
6. ANC ≥1.0 x 109/L, hemoglobin ≥8 g/dL, platelet count ≥75 x 109/L.
7. Calculated creatinine clearance (by Cockroft-Gault) ≥50 mL/min (this equation is as follows: Creatinine clearance in ml/min: (140 - age) x body weight (kg) / 72 x plasma creatinine (mg/dL); multiplied by 0.85 for women) or serum creatinine below 2 g/dL.
8. Negative pregnancy test (serum βHCG) for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 24 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential.
9. FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the study.
10. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
11. Voluntary written informed consent.

Exclusion Criteria:

1. Potential subjects with evidence of progressive disease (CRAB symptoms) as per IMWG criteria.
2. Patient with SPR - significant paraprotein relapse defined as doubling of the M-component in two consecutive measurements separated by < 2 months; or an increase in the absolute levels of serum M protein by 1g/dl, or urine M protein by 500mg /24h, or involved serum FLC level by 20mg/dl (plus an abnormal FLC ratio) in two consecutive measurements separated by < 2 months.
3. Patients who have already started or received post-transplant maintenance or consolidation treatment.
4. Subject has received daratumumab or other anti-CD38 therapies previously.
5. Patients not able to tolerate daratumumab or required concomitant medication and procedures.
6. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
7. Known moderate or severe persistent asthma, or a history of asthma within the last 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study).
8. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
9. Plasma cell leukemia.
10. Waldenström's macroglobulinemia.
11. CNS involvement.
12. Pregnant or lactating females.
13. Radiotherapy within 14 days before randomization. Seven days may be considered if to single area.
14. Major surgery within 3 weeks prior to first dose. Kyfoplasty is not considered as a major surgery.
15. Myocardial infarction within 3 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
16. Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12-lead ECG during screening.
17. Patient who in investigator's opinion is unable to comply with the protocol requirements.
18. Uncontrolled hypertension or diabetes.
19. Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to enter the study.
20. Active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
21. Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone.
22. Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

PREDATOR-MRD:

Inclusion Criteria:

1. Patients with diagnosed symptomatic MM who have completed one or two prior lines of therapy; single or tandem autologous stem cell transplant is not considered a separate line of therapy and is not mandatory; and have achieved CR with negative MRD to the last line of therapy and who remain in CR MRD negative. The last response assessment confirming CR MRD negative status based on assessment of bone marrow sample using flow cytometry with sensitivity of at least 10-5 needs to be performed not earlier than 3 months before inclusion to the study.
2. Males and females ≥18 years of age.
3. Life expectancy of more than 3 months.
4. ECOG performance status of 0-2.
5. Adequate hepatic function, with bilirubin ≤1.5 x ULN and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN.
6. ANC ≥1.0 x 109/L, hemoglobin ≥8 g/dL, platelet count ≥75 x 109/L.
7. Calculated creatinine clearance (by Cockroft-Gault) ≥50 mL/min (this equation is as follows: Creatinine clearance in ml/min: (140 - age) x body weight (kg) / 72 x plasma creatinine (mg/dL); multiplied by 0.85 for women) or serum creatinine below 2 g/dL.
8. Negative pregnancy test (serum βHCG) for women of childbearing potential (including pre-menopausal women who have had a tubal ligation) and for all women not meeting the definition of postmenopausal (≥ 24 months of amenorrhea), and who have not undergone surgical sterilization with a hysterectomy and/or bilateral oophorectomy. For all other women, documentation must be present in medical history confirming that the patient is not of childbearing potential
9. FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the study.
10. Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy.
11. Voluntary written informed consent.

Exclusion criteria:

1. Potential subjects with evidence of progressive disease (CRAB symptoms) as per IMWG criteria.
2. Patient with SPR - significant paraprotein relapse defined as doubling of the M-component in two consecutive measurements separated by < 2 months; or an increase in the absolute levels of serum M protein by 1g/dl, or urine M protein by 500mg /24h, or involved serum FLC level by 20mg/dl (plus an abnormal FLC ratio) in two consecutive measurements separated by < 2 months.
3. Patients who have already started or received post-transplant maintenance or consolidation treatment.
4. Subject has received daratumumab or other anti-CD38 therapies previously.
5. Patients not able to tolerate daratumumab or required concomitant medication and procedures.
6. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
7. Known moderate or severe persistent asthma, or a history of asthma within the last 2 years, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study).
8. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
9. Plasma cell leukemia.
10. Waldenström's macroglobulinemia.
11. CNS involvement.
12. Pregnant or lactating females.
13. Radiotherapy within 14 days before randomization. Seven days may be considered if to single area.
14. Major surgery within 3 weeks prior to first dose. Kyfoplasty is not considered as a major surgery.
15. Myocardial infarction within 3 months prior to enrollment, NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
16. Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12- lead ECG during screening.
17. Patient who in investigator's opinion is unable to comply with the protocol requirements.
18. Uncontrolled hypertension or diabetes.
19. Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to enter the study.
20. Active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
21. Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone.
22. Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Event Free Survival (ESF) | from randomization till the date of development clinical relapse or death from any cause; up to 129 weeks
  To compare (EFS) between daratumumab arm and observation arm after randomization of patients with biochemical relapse of Multiple Myeloma and MRD reappearance in Multiple Myeloma

SECONDARY OUTCOMES:
Overall Response Rate | from randomization till progression or death from any cause, up to 129 weeks
  ORR as determined by Investigator evaluation, defined as the percentage of subjects achieving an objective response (i.e. partial response or better), using IMWG Consensus Panel 1 response criteria
Overall Survival | throughout the duration of the study, no longer than 6 years
  To compare overall survival between arms

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Jamroziak, MD, PhD, Principal Investigator — Polish Myeloma Consortium
Locations (2):
- Poland (2):
  - Szpital Kliniczny Przemienienia Pańskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu; Oddział Hematologii i Transplantacji Szpiku, Poznan, Greater Poland Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: No